CLINICAL TRIAL: NCT02397876
Title: Partially Hydrolyzed Whey Formula in Cow's Milk Allergic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GCO 14-2009
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Food Allergy
Keywords: Food Allergy; Cows Milk Allergy
MeSH Terms: conditions — Food Hypersensitivity; Milk Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- partially hydrolyzed whey formula (Experimental): The group of patients who pass an oral food challenge to partially hydrolyzed whey formula and will be continued on it through out the study
  Interventions: Other: Partially Hydrolyzed Whey formula
- No intervention (No Intervention): Patients who do not pass an oral food challenge to partially hydrolyzed whey formula will continue on their prior diet of cows milk avoidance.

INTERVENTIONS:
Other: Partially Hydrolyzed Whey formula — Patients who tolerate partially hydrolyzed whey formula will be continued on this formula for two years. Patients who do not tolerate the formula will be continued on their prior diet of cows milk avoidance.
  Other Names: Gerber Good Start Formula
  Arms: partially hydrolyzed whey formula

SUMMARY:
Cow's milk (CM) allergy is the most common food allergy in children, affecting 2-3% of infants. In formula-fed infants with CM allergy, extensively hydrolyzed or amino acid-based infant formulas are typically recommended. These formulas are expensive and not palatable. For older patients with CM allergy, the standard of care is avoidance of all CM products. The investigators cared for a CM allergic patient who was able to tolerate partially hydrolyzed whey formula (pHWF), which tastes better and is less expensive than extensively hydrolyzed or amino-acid based formulas. There are likely other subjects who could similarly tolerate pHWF. Furthermore, it is possible that taking pHWF could accelerate tolerance of CM. The investigators aim to identify characteristics of CM allergic subjects who can tolerate pHWF and assess the degree to which taking pHWF accelerates CM tolerance.

DETAILED DESCRIPTION:
Specifically, subjects who have CM allergy will be enrolled. The investigators will perform an oral food challenge (OFC) to pHWF in each subject. Subjects who pass the challenge will be placed on pHWF for 2 years. Subjects who do not pass the challenge will receive routine care. The investigators will perform allergy skin testing, specific IgE measurement, other serologic assays, and longitudinal OFCs to profile subject characteristics in the two groups at baseline and over time.

ELIGIBILITY:
Inclusion Criteria:

* age 0.5-18 years old
* positive skin prick tests (SPT) or detectable serum milk specific IgE and a history of an allergic reaction to milk within 6 months before study screening; or milk-specific IgE level or SPT highly predictive for clinical reactivity (if ≤ 2 years old, sIgE >2 kU/L; if > 2 years old, a level >5 kU/L; SPT wheal diameter ≥ 3 mm)
* a clinical reaction during the cows milk oral food challenge

Exclusion Criteria:

* negative SPT and undetectable milk-specific sIgE
* unstable asthma, allergic rhinitis, or atopic dermatitis
* milk-induced eosinophilic gastroenteropathy
* recent reaction to partially hydrolyzed whey formula
* history of severe anaphylaxis with hypotension to cows milk
* participation in any interventional study for the treatment of food allergy in the 6 months prior to screening visit
* inhalant allergent immunotherapy that has not yet reached maintenance dosing
* inability to discontinue antihistamines for skin testing, OFC
* any systemic therapy which in the judgment of the investigator could be immunomodulatory in the 12 months prior to visit 1 (xolair, rituximab, chronic steroids, etc)
* investigational drug use 90 days prior to visit 1 or intention to use during study period
* the presence of any medical condition that the investigator deems incompatible with participation in the trial.
* unable to understand and speak English

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of partially hydrolyzed whey formula tolerance | Day 1
  Prevalence of partially hydrolyzed whey formula tolerance in cow's milk allergic patients - Identify patients who are cow's milk allergic but can tolerate a partially hydrolyzed whey formula

SECONDARY OUTCOMES:
Time to resolution of cows milk allergy | up to 2 years
  Determine if ingestion of partially hydrolyzed whey formula accelerates the resolution of allergy to cow's milk.

CONTACTS AND LOCATIONS:
Overall Officials: Supinda Bunyavanich, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Wood RA, Sicherer SH, Vickery BP, Jones SM, Liu AH, Fleischer DM, Henning AK, Mayer L, Burks AW, Grishin A, Stablein D, Sampson HA. The natural history of milk allergy in an observational cohort. J Allergy Clin Immunol. 2013 Mar;131(3):805-12. doi: 10.1016/j.jaci.2012.10.060. Epub 2012 Dec 28. PMID 23273958
- [Background] Jin YT. [Surgical treatment of post-traumatic enophthalmos (report of 5 cases)]. Zhonghua Zheng Xing Shao Shang Wai Ke Za Zhi. 1987 Sep;3(3):184-6, 238. No abstract available. Chinese. PMID 3151608
- [Background] Reed RJ, Hairston MA, Palomeque FE. The histologic identity of adenoma sebaceum and solitary melanocytic angiofibroma. Dermatol Int. 1966 Jan-Mar;5(1):3-11. doi: 10.1111/j.1365-4362.1966.tb05174.x. No abstract available. PMID 4293047
- [Background] Lee TD, Gimenez G, Grishina G, Mishoe M, Sampson HA, Bunyavanich S. Profile of a milk-allergic patient who tolerated partially hydrolyzed whey formula. J Allergy Clin Immunol Pract. 2015 Jan-Feb;3(1):116-8. doi: 10.1016/j.jaip.2014.06.021. Epub 2014 Aug 29. No abstract available. PMID 25577632